CLINICAL TRIAL: NCT03946085
Title: Clinical Evaluation of a Micronized, Lipid-based Carotenoid Supplement in Eyes With Retinal Drusen
Brief Title: Evaluation of a New Eye-specific Multivitamin Formula in Participants at Risk of Age-related Macular Degeneration (AMD)
Acronym: AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guardion Health Sciences, Inc. (Industry)
Collaborators: Western University of Health Sciences (Other); Eye Clinic of Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Protocol Number 2
Record Dates: First submitted 2019-04-19; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Retinal Drusen; Age-related Macular Degeneration; Macular Degeneration
Keywords: Lumega-Z; Carotenoid supplement
MeSH Terms: conditions — Retinal Drusen; Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Parallel treatment group participants will be randomly assigned either the experimental intervention, Lumega-Z, or the AREDS2 supplement. An observational, control group will be included for further comparison.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lumega-Z group (Experimental): Participants assigned the study supplement Lumega-Z.
  Interventions: Dietary Supplement: Lumega-Z
- AREDS2 group (Active Comparator): Participants assigned the AREDS2 supplement
  Interventions: Dietary Supplement: AREDS2
- Control (No Intervention): Participants are determined ocular normal after clinical examination and do not have retinal drusen.

INTERVENTIONS:
Dietary Supplement: Lumega-Z — A specially-formulated carotenoid supplement formula that utilizes a micronized, lipid-based liquid form of delivery.
  Other Names: LMZ
  Arms: Lumega-Z group
Dietary Supplement: AREDS2 — A commercially-available multivitamin soft gel formula.
  Other Names: Preservision Age-Related Eye Disease Study 2 (AREDS2)
  Arms: AREDS2 group

SUMMARY:
The aim of this study is to evaluate the clinical benefits in visual function from dietary supplementation of the Lumega-Z carotenoid liquid-supplement in participants with drusen and at risk of AMD. The effects of Lumega-Z supplementation will be compared to an active comparator, the AREDS2 multivitamin.

ELIGIBILITY:
Inclusion Criteria:

- patients with retinal drusen (as determined by clinical fundus photography examination) and dark adaptation recovery time of 6 to 10 minutes.

Exclusion Criteria:

* presence of congenital retinal pathologies that may impact data collection
* prior history of retinal-detachment or vitreo-retinal surgeries with any complications
* best-corrected visual acuity of 20/40 or worse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Mean Changes in Visual Acuity (VA) | Baseline, 3-months, and 6-months
  Repeated measures were obtained using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart-based acuity exam. The ETDRS chart allows a geometric quantification the participant's visual acuity threshold for images under daylight-conditions of black & white contrast. Participant scores were reported as Logarithm of the Minimum Angle of Resolution (LogMAR) units; a more accurate, standardized value equated from the similar acuity charts. Per the clinical evaluation protocol, LogMAR scores of 0.00 - 0.20 are considered "good/normal visual acuity scores"; total range of 0.00 - 1.00. Scores are reported as averaged values, according to each respective group of participants and time-point from which the measurements were collected (i.e. baseline, 3-months, etc...).
  Exclusion criteria included LogMAR scores greater than, or equal to, 0.30 (equivalent to visual acuity of 20/40 or worse).
Mean Changes in Contrast Sensitivity (CS) | Baseline, 3-months, and 6-months
  Contrast Sensitivity Function (CSF) was measured using the CSV-1000E device and measurements were analyzed as logCS units (logarithm of Contrast Sensitivity). The device measures both high- and low-contrast sensitivity (participant's ability to discern size and contrast) within a detection task, and reported as a response-curve. The curve compares the lowest contrast-level for a specific-sized target (across four spatial frequencies; per the manufacturer). Thus, the logCS unit of Contrast Sensitivity, is inversely related to the target's contrast level (displayed by the device). All measurements are reported as averaged values within each group, according to their respective time-frame within the study.
  Normal LogCS scores for adults aged 50-75 years old, in ascending order of spatial frequency (3, 6, 12, and 18), are (1.56 +/- 0.15), (1.80 +/- 0.165), (1.50 +/- 0.15), and (0.93 +/- 0.25). Values were utilized for scale, as recommended by the manufacturer/protocol.
Mean Changes in Dark Adaptation Recovery (DAR) | Baseline, 3-months, and 6-months
  DAR measurements were collected using the AdaptDx adaptometer, to identify the participant's impaired dark adaptation threshold value (in response to low-light condition sensitivity). The device's software reported each patient's sensitivity-value over units of time (minutes), and were recorded as units of Rod Intercept Time. Similarly, measurements reported from each group were an averaged value amongst participant groups at each time-point of collection.
  According to the manufacturing protocol, a Rod Intercept Time of 6.5 minutes was determined to be the cut-off value for part of the inclusion criteria into treatment groups. Previous studies have demonstrated that scores equal to, or greater than, 6.5 minutes are indicative of early-AMD, and those less than 6.5 minutes are considered normal Rod Intercept values.
Mean Changes in Macular Pigment Optical Density (MPOD) | Baseline, 3-months, and 6-months
  MPOD levels were measured by heterochromatic flicker photometry, using the MapCatSF device. MPOD (Macular Pigment Optical Density) measurements represent the level of light absorption by the macular pigment within the central retina, and provide measurements related to macular carotenoid densities. Measurements were reported as LogMAR units (total range of 0.00 to 1.00), as determined by the manufacture software program. Averaged values were reported within each group, at each time-point of collection.
  MPOD values between 0.22 - 0.44 logMAR units have been determined to be middle-range MPOD levels; average value in the USA approximately 0.35. Measurements between (0.0 - 0.21) were considered low-MPOD levels, and those between (0.45 - 1.0) were considered high-MPOD levels. All ranged-scores were obtained by recommendation from the manufacturer.

CONTACTS AND LOCATIONS:
Overall Officials: T Henderson, Principal Investigator — Eye Clinic of Austin
Locations (1):
- Eye Clinic of Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD underlying the results in a publication

REFERENCES:
- [Derived] Davey PG, Henderson T, Lem DW, Weis R, Amonoo-Monney S, Evans DW. Visual Function and Macular Carotenoid Changes in Eyes with Retinal Drusen-An Open Label Randomized Controlled Trial to Compare a Micronized Lipid-Based Carotenoid Liquid Supplementation and AREDS-2 Formula. Nutrients. 2020 Oct 26;12(11):3271. doi: 10.3390/nu12113271. PMID 33114566
- See also: Link to the Lumega-Z medical food — https://lumegaz.com

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT03946085/Prot_SAP_ICF_000.pdf